CLINICAL TRIAL: NCT01197261
Title: An Exploratory, Randomised, Double-blind, Placebo-controlled, Parallel Group, Pilot Study to Assess the Analgesic Efficacy of Oxycodone/Naloxone Prolonged Release Tablets (OXN PR) Compared to Placebo in Opioid-naive Subjects Suffering From Severe Pain Due to Bladder Pain Syndrome.
Brief Title: OXN PR vs Placebo in Opioid-naive Subjects Suffering From Severe Pain Due to Bladder Pain Syndrome (BPS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN2503; 2009-018118-21 (EudraCT Number)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome; Pain
Keywords: Severe pain; Bladder Pain Syndrome; Interstitial Cystitis; Painful Bladder Syndrome; Severe pain due to Bladder Pain Syndrome/Interstitial Cystitis/Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OXN PR (Active Comparator): Oxycodone Naloxone tablets
  Interventions: Drug: Oxycodone naloxone prolonged release tablets
- PLA (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Oxycodone naloxone prolonged release tablets — 2 tablets/ day
  Arms: OXN PR
Drug: Placebo tablets — 2 tablets/ day
  Arms: PLA

SUMMARY:
The study compares the analgesic efficacy of OXN PR vs placebo in opioid-naive subjects suffering from severe pain due to Bladder Pain Syndrome.

DETAILED DESCRIPTION:
The study consists of a screening period followed by randomisation of the patients in a 1:1 ratio to OXN PR treatment or placebo treatment in a double blind fashion. The double blind phase will last for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of severe pain due to Bladder Pain Syndrome (BPS) for at least 6 months
* Subject's treatment of pain due to BPS is insufficient
* Subjects must not have received opioid containing medication in the last 6 months

Exclusion Criteria:

* Females who are pregnant or lactating
* Subjects with any contraindication/history of hypersensitivity to oxycodone, naloxone, paracetamol, related products or other ingredients
* Subjects with any situation in which opioids are contraindicated like severe respiratory depression with hypoxia and/or hypercapnia, severe chronic obstructive lung disease, cor pulmonale, severe bronchial asthma or paralytic ileus
* Evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal or psychiatric disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination that would place the subject at risk upon exposure to the study medication or that may confound the analysis and/or interpretation of the study results
* Abnormal aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatise levels (> 3 times the upper limit of normal), gamma glutamyl transpeptidase > 3 times the upper limit of normal
* Abnormal total bilirubin and/or creatinine level(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To estimate the patient's average pain during treatment with OXN PR compared with placebo | 8 weeks

SECONDARY OUTCOMES:
Patient questionnaires | 8 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Prague, Czechia
- Frankfurt, Germany
- Budapest, Hungary
- Krakow, Poland
- Royal Hallamshire Hospital, Sheffield, United Kingdom

REFERENCES:
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN2503